CLINICAL TRIAL: NCT02821949
Title: Evaluation of Serum Procalcitonin Rate in Patients With Stage IV Non-small Cell Lung
Brief Title: Evaluation of Serum Procalcitonin Rate in Patients With Stage IV Non-small Cell Lung Cancer in First Line Chemotherapy
Acronym: KBPCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2014_843_0012
Record Dates: First submitted 2015-04-10; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Non Small Cells Lung Cancer
Keywords: Non Small Cells Lung Cancer; Procalcitonin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with Non Small Cells Lung Cancer PCT dosage
  Interventions: Biological: PCT dosage

INTERVENTIONS:
Biological: PCT dosage — When connecting chemotherapy products, a PCT dosage will be made. The results of dosage won't be communicated to the clinician responsible for the patient. Patient's care will then be identical to any other chemotherapy treated patient

SUMMARY:
Treatment of a stage IV NSCLC is based on chemotherapy and requires before each session to check clinically, biologically and radiologically absence of infection. This biological evaluation is based on the CRP rate. Lots of infections may occur in this situation and could reduce by three the patient's life duration. However it is very important to make as early as possible a correct diagnosis of infection. CRP rate is classically higher for those patients even without any infection. In comparison with CRP, Procalcitonin (PCT) is well-known for its better sensibility and specificity for the infection diagnosis but has never been study in case of active cancer. The aim of this study is to evaluate the Procalcitonin basal rate for those patients suffering from NSCLC. It could be a simple and reliable method to use. So the investigators decided to include each new patient with NSCLC stage IV coming for his first-line chemotherapy without any infection sign, and to realize a Procalcitonin dosage before the start of the treatment. This sample will be analyzed at the chemical laboratory and the result will not be communicated to the patient physician. A new clinical evaluation will be realized either at the hospital or by phone at day 7 to search any sign of infection. In absence of infection, patient will be reevaluated at day 14, 21 and 30. In case of infection, a new Procalcitonin (and CRP) dosage will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stage IV NSCLC, hospitalized for his first seance of chemotherapy
* Medical conditions permitting chemotherapy
* Informed consent signed
* Patient covered by social insurance

Exclusion Criteria:

* Patient with small cell lung cancer
* Patients with NSCLC stage I, II or III of the Tumor Node Metastasis classification
* Patient with stage IV NSCLC, who received prior treatment (radiotherapy, chemotherapy ...)
* Patient with infection (on clinical and paraclinical criteria) not compatible with the administration of the first seance of chemotherapy.
* Pregnant or breastfeeding women Private Patient freedom or in a position to judicial protection (guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from a stage 4 NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
PCT value performed just before the first chemotherapy treatment | Day 1
  Sampling at the first chemotherapy and each infection

CONTACTS AND LOCATIONS:
Overall Officials: Claire ANDREJAK, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France